CLINICAL TRIAL: NCT05620459
Title: Computer Guided Simultaneous Implant Placement With Ridge Augmentation Using Autogenous Bone Ring Transplant in Defective Maxillary Anterior Sockets
Brief Title: Anterior Maxilla Augmentation Using Chin Bone Ring With Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Gad Mohamed Gad, principal investigator (Master of science student oral and maxillofacial surgery), Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10722
Record Dates: First submitted 2022-11-07; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Ridge Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Ridge augmentation with simultaneous implant placement) (Experimental): Chin bone ring is harvested using surgical guide to augment
  1. anterior maxillary defective recent extraction sockets OR
  2. remaining roots that need extraction and are accompanied with labial bone loss Associated with simultaneous implant placement with the aid of surgical guides
  Interventions: Procedure: Ridge augmentation using chin bone ring with simultaneous implant placement

INTERVENTIONS:
Procedure: Ridge augmentation using chin bone ring with simultaneous implant placement — surgical guides are to be used to harvest chin bone ring, the rings are to be used for bone augmentation in extraction sockets (salama and salama classsification type II),simultaneously implant placement.

SUMMARY:
The study aims toward using autogenous bone grafts to solve decreased bone quantity in anterior maxilla while allowing the patient to recieve implants simultaneously (same time of grafting).

DETAILED DESCRIPTION:
* Chin bone ring will be harvested from patient's(10 in number) chin to augment the recent extraction socket with buccal bone defect, followed by implant placement.
* The process of harvesting and placement of ring will be computer guided which adds lots of accuracy to the bone ring required size from the donor site and the proper placement of both the ring and the implant at the recipient site

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable teeth in the maxillary anterior region with insufficient buccal bone height or buccal bone defect.
* Patients who have given their consent for this trial.
* Both genders males and females will be included.

Exclusion Criteria:

* • Untreated periodontitis.

  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Bone quantity (crestal bone) height) | 3 months after operation day
  Cone beam

SECONDARY OUTCOMES:
Bone quality (bone density at the ring alveolus interface) | 3 months after operation day
  In Hounsfield units making use of ROI region of intrest tool included in the software

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M gad, bds, Principal Investigator — Cairo University
Locations (1):
- cairo University, Cairo, cairo/Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuce MO, Adali E, Turk G, Isik G, Gunbay T. Three-dimensional bone grafting in dental implantology using autogenous bone ring transplant: Clinical outcomes of a one-stage technique. Niger J Clin Pract. 2019 Jul;22(7):977-981. doi: 10.4103/njcp.njcp_652_18. PMID 31293264
- [Background] Omara M, Abdelwahed N, Ahmed M, Hindy M. Simultaneous implant placement with ridge augmentation using an autogenous bone ring transplant. Int J Oral Maxillofac Surg. 2016 Apr;45(4):535-44. doi: 10.1016/j.ijom.2015.11.001. Epub 2015 Nov 28. PMID 26644216
- [Background] Simpson KT, Bryington M, Agusto M, Harper M, Salman A, Schincaglia GP. Computer-Guided Surgery Using Human Allogenic Bone Ring With Simultaneous Implant Placement: A Case Report. Clin Adv Periodontics. 2020 Mar;10(1):16-22. doi: 10.1002/cap.10073. Epub 2019 Oct 14. PMID 31513341
- [Background] Stevens MR, Emam HA, Alaily ME, Sharawy M. Implant bone rings. One-stage three-dimensional bone transplant technique: a case report. J Oral Implantol. 2010;36(1):69-74. doi: 10.1563/AAID-JOI-D-09-00029. PMID 20218871